CLINICAL TRIAL: NCT01923142
Title: Double Blind Within-Subject Controlled Study of Autologous Hair Follicle Outer-Root-Sheath Melanocytes Transplantation in the Treatment of Vitiligo
Brief Title: Efficacy of Autologous Outer-Root-Sheath Melanocytes Transplantation in the Treatment of Vitiligo
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Centro Studi Gised (Other)
Collaborators: ARIV Onlus (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VIT-FOL1
Record Dates: First submitted 2013-08-09; First posted 2013-08-15 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Vitiligo
Keywords: Vitiligo; Outer-Root-Sheath; Melanocytes; Hair Follicles
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Outer-Root-Sheath Melanocytes Suspension (Experimental): This arm includes all patients sides (left or right) treated with autologous outer-root-sheath melanocytes suspension followed by targeted UVB phototherapy
  Interventions: Biological: Outer-Root-Sheath Melanocytes Suspension
- Placebo (Placebo Comparator): This arm includes all patients sides (left or right) treated with placebo followed by targeted UVB phototherapy
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Outer-Root-Sheath Melanocytes Suspension — The treatment consists in depositing a suspension of autologous outer-root-sheath melanocytes, derived from patient's plucked hair follicles, and patient's own serum on the area affected by vitiligo, after properly preparation with dermabrasion. Afterwards a targeted UVB phototherapy will be carried out by patients at home for 3 days / week from the beginning of the 5th week after transplantation till the end of the study period (12th week).
  Arms: Outer-Root-Sheath Melanocytes Suspension
Biological: Placebo — The treatment consists in depositing a solution made of saline and patient's own serum on the area affected by vitiligo, after properly preparation with dermabrasion. Afterwards a targeted UVB phototherapy will be carried out by patients at home for 3 days / week from the beginning of the 5th week after transplantation till the end of the study period (12th week).
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the hypothesis that, in patients with stable vitiligo unresponsive to conventional treatments including traditional phototherapy and/or topical steroids, the application of a non-cultured autologous hair follicle outer-root-sheath melanocytes suspension in the area affected by the disease followed by targeted ultraviolet B (UVB) phototherapy can lead to a significant skin repigmentation. To assess the effect of the proposed treatment, a within-subject controlled study involving selected symmetric lesion areas localized to the back of the hands will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Presence of symmetric lesions of vitiligo at the back of the hands with an extension >5cm²
* Vitiligo lasting at least one year at the backs of both hands
* Stable vitiligo, defined as vitiligo that presents no evident evolution (appearance of new lesions or increase in the extension of lesions already present) for at least 6 months
* Suspension for at least two months prior to the enrollment date of any systemic drug for vitiligo such as immunosuppressive treatment (cyclosporine, systemic steroids) or psoralen + ultraviolet A therapy, phototherapy with ultraviolet B, and of any anticoagulant drug
* Suspension of topical medications for at least 15 days prior to the enrollment date

Exclusion Criteria:

* Presence of active vitiligo or Koebner phenomenon
* Difference of more than 10% in the extension of symmetrical areas of vitiligo
* Presence of systemic infections or infections localized to the tissues intended for transplantation
* History of infections to the tissues intended for transplantation (herpes simplex, human papillomavirus infections, pityriasis versicolor, pityriasis alba)
* Presence or history of malignancy
* Chemotherapy or radiation therapy in progress
* History of allergies or adverse reactions to local anesthetics
* Presence of transmissible diseases (human immunodeficiency virus, hepatitis B and C, human T-lymphotropic virus type I and II, syphilis, cytomegalovirus, Creutzfeldt-Jacob, tuberculosis)
* Women who are pregnant or intend to become pregnant during the study period (including breastfeeding women)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Repigmentation equal to or greater than 50% of the treated areas from baseline as assessed by image analysis | 12 weeks

SECONDARY OUTCOMES:
Any repigmentation of the treated areas from baseline as assessed by physician according to an ordinal 6-points scale | 6 weeks, 12 weeks
Any repigmentation of the treated areas from baseline as assessed by patient according to an ordinal 6-points scale | 6 weeks, 12 weeks
Overall patient satisfaction to the proposed therapy as assessed by visual analogue scale | 6 weeks, 12 weeks
Any repigmentation of the treated areas from baseline as assessed by image analysis | 6 weeks, 12 weeks
Any repigmentation of other areas affected by vitiligo from baseline as assessed by physician according to an ordinal 6-points scale (evaluation of a possible systemic effect) | 6 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Naldi, MD, Principal Investigator — Centro Studi Gised
Locations (2):
- Italy (2):
  - Papa Giovanni XXIII Hospital, Bergamo
  - Spedali Civili, Brescia